CLINICAL TRIAL: NCT03734302
Title: A Single-center, Open-label Study Evaluating the Pharmacokinetics, and Safety of Multiple Dose Oral Brexpiprazole Tablets (1 mg) in Chinese Healthy Subjects
Brief Title: The Pharmacokinetics, and Safety of Brexpiprazole Tablets in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 331-403-00025
Record Dates: First submitted 2018-11-02; First posted 2018-11-07 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple dose oral administration (Experimental): 1mg Once Daily (QD) , oral administration,14 consecutive days
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole , mutiple dose /oral/empty stomach
  Other Names: Brex

SUMMARY:
This study is a single-center, open-label study evaluating the pharmacokinetics and safety of multiple dose oral administration of Brexpiprazole (1 mg) tablets in Chinese healthy subject.10 healthy adult subjects will be enrolled in this study. A single dose (Brexpiprazole 1 mg) group is set and the test drug will be administered for 14 consecutive days.

DETAILED DESCRIPTION:
10 healthy adult subjects will be enrolled in this study. A single dose (Brexpiprazole 1 mg) group is set and the test drug will be administered for 14 consecutive days.

After receiving the informed consent form the subject themselves, the investigators start the screening 14 days to 1 days prior to taking the study drug (D-14 to D-1).

One day before first dosing (D-1), subjects are hospitalized. On the next day (D1), after completed the hospitalization inspection, eligible subjects will be selected to start with the first dose, and from day 1 to day 14 (D1 to D14), continue once daily dosing and complete the corresponding inspection, observation and blood sampling. They continue hospitalization and are discharged on day 17 (D17) after completing the relevant examinations. On days 19, 21, 23，25 (D19, D21，D23 and D25), blood samples are collected and safety evaluation is performed.

Telephone follow-up is performed on day 44 (D44, 30 days after the last dose of the drug).

Subjects who early terminated the test after taking the study drug should be tested at the end of the study (D25/ET) as far as possible.

Blood samples for pharmacokinetic evaluation are collected before daily dosing; D1 (before dosing, and 1, 2, 3, 4, 5, 6, 8, 12 hours after dosing), D2 (before dosing and 24 hours after first dosing), D10 (before dosing), D11 (before dosing), D12 (before dosing), D13 (before dosing), D14 (before dosing, and 1, 2, 3, 4, 5, 6, 8, 12 hours after dosing), D15 (24 hours after last dosing), D16 (48 hours after last dosing), D17 (72 hours after last dosing), D18 (96 hours after last dosing), D19 (120 hours after last dosing), D21 (168 hours after last dosing),D23 (216 hours after last dosing), D25 (264 hours after last dosing). 31 Blood samples collecting points in total.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign the informed consent form
* 2. At the age of 18~45 years old (including upper and lower limits).
* 3. Body weight of not less than 45 kg, body mass index 19 ~ 25kg/m2 range (including the upper and lower limits) [ body mass index (BMI) = body weight (kg) / height2 (m2)].

Exclusion Criteria:

* 1. Participated in any drug test within 12 weeks prior to enrollment.
* 2. Drug abuse in the past 2 years or a history of substance abuse.
* 3. Drinking alcohol more than 2 unit per day (1 unit= 360 ml beer , or 45 ml 4.0% alcohol, or 150 ml liquor, or 50 ml wine ) 6 months before the screening, or subjects can not stop drinking during the hospitalization.
* 4. Drug abuse urine test at screening is positive.

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Steady-state peak time (Tss_max) | Day1, Day2, Day10, Day11, Day12, Day13, Day14, Day15, Day16, Dv17, Day18, Day19, Dv21,Day23, Day25
  Assessment of the steady-state peak time of Brexpiprazole
Steady-state valley concentration(Css_min) | Day1, Day2, Day10, Day11, Day12, Day13, Day14, Day15, Day16, Dv17, Day18, Day19, Dv21,Day23, Day25
  Assessment of the steady-state valley concentration of Brexpiprazole
Steady-state peak concentration (Css_max) | Day1, Day2, Day10, Day11, Day12, Day13, Day14, Day15, Day16, Dv17, Day18, Day19, Dv21,Day23, Day25
  Assessment of the steady-state peak concentration of Brexpiprazole
Average steady-state plasma concentration (Css_av) | Day1, Day2, Day10, Day11, Day12, Day13, Day14, Day15, Day16, Dv17, Day18, Day19, Dv21,Day23, Day25
  Assessment of the average steady-state plasma concentration (Css_av) of Brexpiprazole
Half-life (t1/2, z) | Day1, Day2, Day10, Day11, Day12, Day13, Day14, Day15, Day16, Dv17, Day18, Day19, Dv21,Day23, Day25
  Assessment of the Half-life of Brexpiprazole
Steady-state clearance (CLss/F) | Day1, Day2, Day10, Day11, Day12, Day13, Day14, Day15, Day16, Dv17, Day18, Day19, Dv21,Day23, Day25
  Assessment of the steady-state clearance of Brexpiprazole
Area under steady state plasma concentration-time curve (AUC)ss | Day1, Day2, Day10, Day11, Day12, Day13, Day14, Day15, Day16, Dv17, Day18, Day19, Dv21,Day23, Day25
  Assessment of the area under steady state plasma concentration-time curve of Brexpiprazole
Fluctuation index (DF) | Day1, Day2, Day10, Day11, Day12, Day13, Day14, Day15, Day16, Dv17, Day18, Day19, Dv21,Day23, Day25
  Assessment of the fluctuation index of Brexpiprazole
Cumulative coefficient (RAUC, Rcmax) | Day1, Day2, Day10, Day11, Day12, Day13, Day14, Day15, Day16, Dv17, Day18, Day19, Dv21,Day23, Day25
  Assessment of the cumulative coefficient of Brexpiprazole

SECONDARY OUTCOMES:
The peak concentration (Cmax) after the first administration | Day1, Day2
  The peak concentration (Cmax) of Brexipiprazole and the metabolite DM-3411 on the first day after administration are calculated.
The peak time (Tmax) after the first administration | Day1, Day2
  The peak-time of Brexipiprazole and the metabolite DM-3411 on the first day after administration are calculated.
Area under the plasma concentration-time curve (AUC0-24h) | Day1, Day2
  The area under the plasma concentration-time curve of Brexipiprazole and the metabolite DM-3411 on the first day after administration are calculated.
Valley concentration points | Day10, Day11, Day12, Day13, Day14
  Descriptive statistics about the valley concentration points before taking the study drug on days 10, 11, 12, 13 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, Master, Principal Investigator — Beijing Anding Hospital of Capital Medical University
Locations (1):
- Beijing Anding Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No